CLINICAL TRIAL: NCT02187146
Title: The Effects of Serum Vitamin D and IVF Outcome: a Prospective Cohort Study
Brief Title: The Effects of Serum Vitamin D and IVF Outcome
Acronym: VIDIO
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Responsible Party: Principal Investigator, Justin Chu, Research Fellow, University of Birmingham
Other Study IDs: RG_13-100
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Deficiency; Vitamin D Insufficiency; Infertility
Keywords: Vitamin D; Infertility; IVF; ART
MeSH Terms: conditions — Vitamin D Deficiency; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ART population: Patients undergoing IVF/ICSI/FET treatment at the Birmingham Womens Fertility Centre 2013-2014

SUMMARY:
The purpose of this study is to investigate whether an association exists between serum vitamin D levels and IVF treatment outcome

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing IVF, ICSI or FET treatment at Birmingham Womens Fertility Centre

Exclusion Criteria:

* None

Ages: 23 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients undergoing IVF, ICSI and FET treatment cycles at the Birmingham Womens Fertility Centre
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 7 weeks after embryo transfer
  USS appearances of intrauterine pregnancy

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 2 weeks after embryo transfer
  Urinary pregnancy test result 2 weeks after embryo transfer
Miscarriage rate | 20 weeks after embryo transfer
  Pregnancy outcome of miscarriage
Live birth rate | 42 weeks after embryo transfer
  Live birth outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham Womens NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Chu J, Gallos I, Tobias A, Robinson L, Kirkman-Brown J, Dhillon-Smith R, Harb H, Eapen A, Rajkhowa M, Coomarasamy A. Vitamin D and assisted reproductive treatment outcome: a prospective cohort study. Reprod Health. 2019 Jul 15;16(1):106. doi: 10.1186/s12978-019-0769-7. PMID 31307482